CLINICAL TRIAL: NCT05075772
Title: Absolute Bioavailability, Safety, Tolerability, and Pharmacodynamics Following Subcutaneous (SC) Injection of 100 mg BI 765080 Relative to Intravenous (IV) Dose in Healthy Male Subjects
Brief Title: A Study in Healthy Men to Test How BI 765080 is Taken up in the Body When Given as an Injection Under the Skin Compared With an Infusion Into the Vein
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1450-0002; 2021-003281-13 (EudraCT Number)
Record Dates: First submitted 2021-09-30; First posted 2021-10-13 (Actual); Results first posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-03

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 100 mg BI 765080 SC injection (T) (Experimental)
  Interventions: Drug: BI 765080
- 100 mg BI 765080 IV infusion (R) (Experimental)
  Interventions: Drug: BI 765080

INTERVENTIONS:
Drug: BI 765080 — BI 765080

SUMMARY:
A study in healthy man to investigate the absolute bioavailability of 100mg BI 765080, once administered as subcutaneous (SC) injection and once administered as intravenous infusion.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Caucasian male subjects according to the assessment of the investigator, as based on a complete medical history, a physical examination, vital signs (Blood Pressure (BP), Pulse Rate (PR)), 12- lead Electrocardiogram (ECG), and clinical laboratory tests
* Age of 18 to 55 years (inclusive)
* Body mass index (BMI) of 18.5 to 29.9 kg/m2 (inclusive)
* Signed and dated written informed consent prior to admission to the study, in accordance with Good clinical practice (GCP) and local legislation

Exclusion Criteria:

* Any finding in the medical examination (including ECG) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 millimetre of mercury (mmHg), diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 45 to 90 beats per minute (bpm)
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections Further exclusion criteria apply.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2021-10-25 (Actual); Primary Completion 2022-03-11 (Actual); Study Completion 2022-03-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- SGS Life Science Services - Clinical Research, Edegem, Belgium

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phase 1 to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the licence holder;
  2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials;
  3. studies conducted in a single center or targeting rare disease (because of limitations of anonymization).
  For more details refer to: http://mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — http://mystudywindow.com/msw/datasharing

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was randomized, open-label, and single-dose, with matched parallel groups (test treatment (T) group: subcutaneous (SC) injection of 100 milligram (mg) BI 765080; reference treatment (R) group: intravenous (IV) infusion of 100 mg BI 765080). Subjects in the T and R groups were matched based on age and body weight.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trail. Subjects attend a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- 100 mg BI 765080 SC Injection (T): Participants were administered a single dose of 100 milligram (mg) of BI 765080 as subcutaneous injection (SC).
- 100 mg BI 765080 IV Infusion (R): Participants were administered a single dose of 100 milligram (mg) of BI 765080 as intravenous infusion (IV).
Period: Overall Study
Arm/Group | 100 mg BI 765080 SC Injection (T) | 100 mg BI 765080 IV Infusion (R)
Started | 14 | 14
Completed | 14 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated Set: Included all subjects who were randomised and treated with a dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | 100 mg BI 765080 SC Injection (T) | 100 mg BI 765080 IV Infusion (R) | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.4 (12.2) | 41.1 (10.3) | 40.8 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 14 | 14 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 14 | 14 | 28
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 14 | 14 | 28
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 81.91 (9.72) | 82.92 (9.01) | 82.41 (9.21)

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve of BI 765080 in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point (AUC0-tz)
Description: Area under the concentration-time curve of BI 765080 in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz) is reported.
Time Frame: Within 3 hours (h) before and 0.5h, 2h, 4h, 8h, 12h, 24h, 34h, 48h, 72h, 96h*, 120h, 168h, 240h, 312h, 480h, 648h and 1320h after administration of BI 765080. * Applicable only for the arm "100 mg BI 765080 SC injection (T)"
Population: The pharmacokinetic (PK) parameter analysis set (PKS): Including all subjects in the treated set (TS) who provided non-excluded data for at least one primary or secondary PK endpoint. Descriptive and model-based analyses of PK parameters were based on the PKS.
Measure: Geometric Least Squares Mean (Standard Error); unit: hours*nanogram/milliliter
Arm/Group | 100 mg BI 765080 SC Injection (T) | 100 mg BI 765080 IV Infusion (R)
Number analyzed (Participants) | 13 | 14
hours*nanogram/milliliter | 3528304.5 (NA) — Adjusted geometric standard error= 1.082 | 7625263.8 (NA) — Adjusted geometric standard error= 1.079
Statistical Analysis 1: Comparison: 100 mg BI 765080 SC Injection (T) vs 100 mg BI 765080 IV Infusion (R); The statistical model used for the analysis of this primary endpoint was an analysis of variance (ANOVA). The PK endpoints were log-transformed (natural logarithm) prior to fitting the ANOVA model. The model included a fixed effect for treatment assignment and a random effect for matching pair (each matched pair in the study was assigned a number for the analysis); Test type: Other; Ratio of gMeans (%) = 46.3, 90% CI 2-sided [38.3 to 55.9] — Ratio of Geometric Least Squares Means (gMeans) was calculated as (gMean of "SC injection (T)")/(gMean of "IV infusion (R)"). Intra-matched-pair geometric coefficient of variation=28.2

2. Primary Outcome: Maximum Measured Concentration of BI 765080 in Plasma (Cmax)
Description: Maximum measured concentration of BI 765080 in plasma (Cmax) is reported.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Least Squares Mean (Standard Error); unit: nanogram/milliliter
Arm/Group | 100 mg BI 765080 SC Injection (T) | 100 mg BI 765080 IV Infusion (R)
Number analyzed (Participants) | 13 | 14
nanogram/milliliter | 9582.0 (NA) — Adjusted geometric standard error= 1.064 | 35718.4 (NA) — Adjusted geometric standard error= 1.061
Statistical Analysis 1: Comparison: 100 mg BI 765080 SC Injection (T) vs 100 mg BI 765080 IV Infusion (R); [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratio of gMeans (%) = 26.8, 90% CI 2-sided [23.2 to 31.1] — Ratio of Geometric Least Squares Means (gMeans) was calculated as (gMean of "SC injection (T)")/(gMean of "IV infusion (R)"). Intra-matched-pair geometric coefficient of variation=22.5

3. Secondary Outcome: Area Under the Concentration-time Curve of the Analyte in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞)
Description: Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞) is reported.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Least Squares Mean (Standard Error); unit: hours*nanogram/milliliter
Arm/Group | 100 mg BI 765080 SC Injection (T) | 100 mg BI 765080 IV Infusion (R)
Number analyzed (Participants) | 13 | 14
hours*nanogram/milliliter | 3590175.4 (NA) — Adjusted geometric standard error= 1.080 | 7638615.9 (NA) — Adjusted geometric standard error= 1.077
Statistical Analysis 1: Comparison: 100 mg BI 765080 SC Injection (T) vs 100 mg BI 765080 IV Infusion (R); The statistical model used for the analysis of this secondary endpoint was an analysis of variance (ANOVA). The PK endpoints were log-transformed (natural logarithm) prior to fitting the ANOVA model. The model included a fixed effect for treatment assignment and a random effect for matching pair (each matched pair in the study was assigned a number for the analysis); Test type: Other; Ratio of gMeans (%) = 47.0, 90% CI 2-sided [39.0 to 56.6] — Ratio of Geometric Least Squares Means (gMeans) was calculated as (gMean of "SC injection (T)")/(gMean of "IV infusion (R)"). Intra-matched-pair geometric coefficient of variation=27.7

4. Secondary Outcome: Occurrence of Drug-related Adverse Events
Description: Percentage of participants with drug-related adverse events is reported.
Time Frame: From start of drug of administration until end of trial, up to 59 days.
Population: Treated Set: Included all subjects who were randomised and treated with a dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | 100 mg BI 765080 SC Injection (T) | 100 mg BI 765080 IV Infusion (R)
Number analyzed (Participants) | 14 | 14
percentage of participants | 28.6 | 7.1

ADVERSE EVENTS:
Time Frame: From start of drug of administration until end of trial, up to 59 days.
Description: Treated Set: Included all subjects who were randomised and treated with a dose of study drug.
Arm/Group | 100 mg BI 765080 SC Injection (T) | 100 mg BI 765080 IV Infusion (R)
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 8/14 | 2/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 100 mg BI 765080 SC Injection (T) (N=14) | 100 mg BI 765080 IV Infusion (R) (N=14)
Injection site reaction (General disorders) | 2 | 0
Medical device site irritation (General disorders) | 1 | 0
Sense of oppression (General disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
COVID-19 (Infections and infestations) | 2 | 0
Dizziness (Nervous system disorders) | 0 | 2
Dysgeusia (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Electrocardiogram repolarisation abnormality (Investigations) | 1 | 0
Abnormal dreams (Psychiatric disorders) | 0 | 1
Agitation (Psychiatric disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2021-10-20): https://cdn.clinicaltrials.gov/large-docs/72/NCT05075772/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-08): https://cdn.clinicaltrials.gov/large-docs/72/NCT05075772/SAP_001.pdf